CLINICAL TRIAL: NCT06230523
Title: A Phase 2, Parallel-Group, Double-Blind Study to Investigate Weight Management With LY3841136 Compared With Placebo in Adult Participants With Obesity or Overweight
Brief Title: A Study of LY3841136 Compared With Placebo in Adult Participants With Obesity or Overweight
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18808; W8M-MC-LAA1 (Other: Intervention-specific appendix (ISA) number); CWMM Master Protocol (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Overweight and Obesity
Keywords: Overnutrition; Hormones; Chronic weight management
MeSH Terms: conditions — Obesity; Overweight; Overnutrition

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- LY3841136 Dose 1 (Experimental): Participants will receive LY3841136 subcutaneously (SC)
  Interventions: Drug: LY3841136
- LY3841136 Dose 2 (Experimental): Participants will receive LY3841136 SC
  Interventions: Drug: LY3841136
- LY3841136 Dose 3 (Experimental): Participants will receive LY3841136 SC
  Interventions: Drug: LY3841136
- LY3841136 Dose 4 (Experimental): Participants will receive LY3841136 SC.
  Interventions: Drug: LY3841136
- LY3841136 Dose 5 (Experimental): Participants will receive LY3841136 SC
  Interventions: Drug: LY3841136
- LY3841136 Dose 6 (Experimental): Participants will receive LY3841136 SC
  Interventions: Drug: LY3841136
- Placebo (Placebo Comparator): Participants will receive LY3841136 matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3841136 — Administered SC.
  Arms: LY3841136 Dose 1; LY3841136 Dose 2; LY3841136 Dose 3; LY3841136 Dose 4; LY3841136 Dose 5; LY3841136 Dose 6
Drug: Placebo — Administered SC.
  Arms: Placebo

SUMMARY:
The main purpose of this study, performed under the master protocol W8M-MC-CWMM (NCT06143956), is to investigate weight management efficacy and safety with LY3841136 compared with placebo in adult participants with obesity or overweight. The study will last about 64 weeks and may include up to 17 visits.

ELIGIBILITY:
Inclusion Criteria:

W8M-MC-LAA1

* Are males and females who agree to abide by the reproductive and contraceptive requirements

W8M-MC-CWMM:

* Have a BMI ≥27 kg/m²
* Have had a stable body weight for the 3 months prior to randomization (<5% body weight gain and/or loss)

Exclusion Criteria:

W8M-MC-LAA1

* Have any prior diagnosis of diabetes mellitus except gestational diabetes.
* Have any of the following cardiovascular conditions within 6 months prior to screening:

  * acute myocardial infarction
  * cerebrovascular accident (stroke)
  * unstable angina, or
  * hospitalization due to congestive heart failure (CHF).
* Have a history of acute or chronic pancreatitis.
* Have an on-going or history of bradyarrhythmia and/or sinus bradycardia at screening and baseline.

W8M-MC-CWMM

* Have a prior or planned surgical treatment for obesity, except prior liposuction or abdominoplasty, if performed >1 year prior to screening.
* Have type 1 diabetes mellitus, latent autoimmune diabetes in adults, or history of ketoacidosis or hyperosmolar coma.
* Have poorly controlled hypertension.
* Have a history of symptomatic gallbladder disease within the past 2 years
* Have signs and symptoms of any liver disease other than nonalcoholic fatty liver disease.
* Have a lifetime history of suicide attempts.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 48

SECONDARY OUTCOMES:
Change from Baseline in Body Weight | Baseline, Week 48
Percentage of Participants Who Achieve ≥5% Body Weight Reduction | Baseline to Week 48
Percentage of Participants Who Achieve ≥10% Body Weight Reduction | Baseline to Week 48
Change from Baseline in Body Mass Index (BMI) | Baseline, Week 48
Pharmacokinetics (PK): Area Under the Curve (AUC) of LY3841136 | Baseline to Week 48
PK: Maximum Concentration (Cmax) of LY3841136 | Baseline to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (46):
- United States (43):
  - The Institute for Liver Health II dba Arizona Clinical Trials - Mesa, Chandler, Arizona
  - Headlands Research - Scottsdale, Scottsdale, Arizona
  - The Institute for Liver Health II dba Arizona Liver Health-Tucson, Tucson, Arizona
  - NorCal Medical Research, Inc, Greenbrae, California
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Northeast Research Institute (NERI), Fleming Island, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Charter Research - Winter Park, Orlando, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Pacific Diabetes & Endocrine Center, Honolulu, Hawaii
  - Medical Research Partners, Ammon, Idaho
  - Great Lakes Clinical Trials - Andersonville, Chicago, Illinois
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - NorthShore University Health System, Skokie, Illinois
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Knownwell, Needham, Massachusetts
  - Lucida Clinical Trials, New Bedford, Massachusetts
  - Headlands Research - Detroit, Southfield, Michigan
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Dent Neurologic Institute, Amherst, New York
  - Velocity Clinical Research, Syracuse, East Syracuse, New York
  - North Suffolk Neurology, Port Jefferson Station, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - Medication Management, Greensboro, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Lucas Research, Inc., New Bern, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Quality Medical Research, Nashville, Tennessee
  - IMA Clinical Research Austin, Austin, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Tekton Research - Fredericksburg Road, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Spectrum Medical, Inc., Danville, Virginia
  - Central Washington Health Services Association d/b/a Confluence Health, Wenatchee, Washington
- Argentina (3):
  - Centro Médico Viamonte, Buenos Aires, Buenos Aires F.D.
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires, Buenos Aires F.D.
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Billings LK, Hsia S, Bays H, Tidemann-Miller B, O'Hagan J, Tham LS, Butler A, Kazda C, Mather KJ, Coskun T. Eloralintide, a selective amylin receptor agonist for the treatment of obesity: a 48-week phase 2, multicentre, double-blind, randomised, placebo-controlled trial. Lancet. 2025 Dec 6;406(10520):2631-2643. doi: 10.1016/S0140-6736(25)02155-5. Epub 2025 Nov 6. PMID 41207310
- See also: A Study of LY3841136 Compared With Placebo in Adult Participants With Obesity or Overweight — https://trials.lilly.com/en-US/trial/454455